CLINICAL TRIAL: NCT06822751
Title: Exploratory Pragmatic Trial of Fosfomycin-trometamol Treatment of Male Urinary Tract Infections in Primary Care
Brief Title: FOsfomycin for Male Urinary Tract Infection
Acronym: FOMUTI
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: INSERM UMR1311 DYNAMICURE (Unknown); Department of General Practice, Rouen University (Unknown); Health Ministry funding (ReSpiR funds) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/0376/HP; 2023-510355-36-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-22; First posted 2025-02-12 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Urinary Tract Infection; Prostatitis; Cystitis
Keywords: Men; Cystitis; Urinary Tract Infection; Anti-infective agents, urinary; Fosfomycin
MeSH Terms: conditions — Urinary Tract Infections; Prostatitis; Cystitis; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- fosfomycine-trometamol (Experimental): Single-Arm The treatment studied is fosfomycin trometamol (FT): FOSFOMYCINE ARROW ADULTS 3 g, granule for drinkable solution in sachet.
  FT is available in generic form. It comes in a sachet of 3 g of granules for oral solution (orange flavour).
  In this study, FT will be taken to treat a non-febrile male urinary tract infection, at a dosage of 3 g per day every 2 days for 14 days, i.e. 7 doses (D0, D2, D4, D6, D8, D10, D14). Seven sachets, accompanied by a prescription specifying the dosage, will therefore be given to the patient on inclusion in the study.
  Interventions: Drug: Fosfomycun-trometamol

INTERVENTIONS:
Drug: Fosfomycun-trometamol — Study of the efficacy and safety of Fosfomycin trometamol as a 14-day treatment using a 3 g sachet every 2 days for 14 days for the treatment of male urinary tract infections in primary care: open-label, non-randomised, multicentre, inter-regional trial.

SUMMARY:
Male urinary tract infections (MUTI) are often less recognised compared to those in women. French clinical guidelines practices recommend the use of antibiotics called fluoroquinolones, which are highly effective in treating MUTIs. However, these antibiotics can lead to rare but serious side effects, such as tendonitis or heart rhythm disturbances. Additionally, fluoroquinolones can contribute to the development of bacterial resistance, making their use inadvisable within six months of treatment.

In response to these concerns, we aim to explore a well-established alternative, fosfomycin trometamol (known by the brand name MONURIL®). This antibiotic has a strong track record in treating UTIs in women, with well-documented benefits and minimal associated risks.

The primary goal of this study is to assess the effectiveness of fosfomycin trometamol in treating urinary tract infections in men, as well as to evaluate any potential treatment failures.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years or older.
* Consulting in a primary care setting.
* Suspected of having a male urinary tract infection (MUTI) by the investigating physician and presenting at least one recent acute symptom (< 3 months) from the following:

  * Lower urinary tract symptoms: dysuria, urgency, frequency, hematuria.
  * Pelvic pain unrelated to urination: suprapubic, perineal, or urethral pain.
* Patient has read and understood the information letter and signed the informed consent form.
* Affiliation with a social security system or beneficiary of such a system.
* No history of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participation in the protocol or to prevent him/her from giving informed consent

Exclusion Criteria:

* Presence of one or more criteria for severity of infection

  * Severe sepsis or septic shock defined by a qSOFA score ≥ 2
  * or/and systolic BP less than 100 mmHg: non-inclusion criterion
  * or/and temperature < 36°C or > 38°C
  * or/and diagnosis of pyelonephritis (pain on lumbar percussion)
  * or/and presence of abdominal guarding/contraction
  * or/and presence of a bladder globe above the pubic bone: (suspected acute retention of urine)
  * or/and known immunosuppression: any immunosuppressive treatment (including corticosteroid therapy > 10 mg/d for more than 5 days), neutropenia (PNN < 500/mL) severe malnutrition (albumin < 30 and/or BMI < 16),
* No diagnosis of male urinary tract infection in the last 3 months,
* No ongoing chronic prostatitis,
* Known urinary tract abnormality: urinary tract lithiasis, vesico-ureteral reflux, prostate or urinary tract cancer, prostate adenoma treated medically or surgically, urinary tract malformation (including single kidney and urethral stricture).
* Acute retention of urine and indication for surgical or interventional drainage
* Hyperalgesic form
* Urinary tract infection associated with care, on urinary catheter or suprapubic catheter
* Urinary tract surgery, cystoscopy, prostate biopsy or urinary catheterisation less than 3 months old
* Urinary tract surgery, cystoscopy, prostate biopsy or urinary catheterisation less than 3 months old
* Severe disease or high probability of death within 3 months,
* Hypersensitivity to fosfomycin trometamol or to any of the excipients (notable excipients: sucrose, dextrose (source of glucose), maltodextrin (source of glucose), orange yellow colouring S (E110)),
* End-stage renal disease (creatinine clearance <10 mL/min),
* Patients with glucose and galactose malabsorption syndrome or sucrase/isomaltase deficiency (rare hereditary disease)
* Antibiotic taken within 72 hours of diagnosis of male urinary tract infection,
* Major cognitive impairment,
* Person deprived of liberty by an administrative or judicial decision or person placed under court protection / sub- guardianship or curatorship
* Any history of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participation in the protocol or to prevent the subject from giving informed consent.
* Known non-adherence to treatment,
* Simultaneous participation in another interventional clinical study,
* Cannot be taken orally (vomiting)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of 14 days of fosfomycin trometamol (FT) treatment for non-febrile male urinary tract infections (MUTIs) in primary care | 14 days
  The primary endpoint was defined as the absence of clinical failure up to 14 days after the end of antibiotic treatment.
  Failure is defined according to SPILF recommendations as :
  * a change of antibiotic treatment to a reference treatment (see above) for urinary tract infection ;
  * and/or hospitalisation for urinary tract infection ;
  * or/and acute retention of urine ;
  * or/and a new consultation for worsening or persistence of symptoms ;
  * or/and the appearance of a fever > 38°C

SECONDARY OUTCOMES:
Nosological (clinical and biological) description of non-febrile male urinary tract infections (MUTIs) managed in primary care. | 3 months
  Improvement in functional urinary symptomatology using a Lickert scale (1. Very unsignificant, 2. Unsignificant , 3. Neither , 4. Significant , 5. Very significant) , 2-5 days 28-35 days and 3 months after the start of treatment with FT;
Clinical cure rate 10 to 12 weeks after inclusion (i.e., 8 to 10 weeks after completion of fosfomycin trometamol (FT) treatment) | 8 to 10 weeks after completion of fosfomycin trometamol (FT) treatment
  cytobacteriological examination of the urine (CBEU) negative 10 to 12 weeks after the end of treatment ;
Microbiological cure rate (assessed by cytobacterial examination of urine), at 14 to 21 days and 10 to 12 weeks after inclusion. | at 14 to 21 days and 10 to 12 weeks after inclusion.
  Negative cytobacteriological examination of the urine (CBEU) (leucocyturia < 10/mm3 OR leucocyturia > 10/mm3 AND bacteriuria < 103/mm3 or bacteriuria with a different pathogen) taken 14 to 21 days after the end of antibiotic treatment
Establishment of a repository of uropathogens responsible for MUTIs. | 3 months
  Regression of urinary signs 10 to 12 weeks after the end of treatment;
Analysis of treatment-related adverse effects, 14 days after inclusion | 14 days after inclusion
  Adverse events presented by the patient and recorded by the investigating doctor during antibiotic treatment and in the 14 days following the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dr SOUDAIS, MD, Principal Investigator — University Rouen Hospital

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD for this study